CLINICAL TRIAL: NCT04505397
Title: A Phase 1, Randomized, Double-Blinded, Single-Dose Escalation Study Followed by a Multiple-Dose Escalation Study of SKL24741 in Healthy Subjects
Brief Title: Single-Dose Escalation Study Followed by a Multiple-Dose Escalation Study of SKL24741 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKL24741C001
Record Dates: First submitted 2020-01-30; First posted 2020-08-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (22):
- Single Ascending Dose Level 1 (Experimental): 4 Subjects will receive one dose of 10 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 2 (Experimental): 4 Subjects will receive one dose of 25 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 3 (Experimental): 4 Subjects will receive one dose of 50 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 4 (Experimental): 4 Subjects will receive one dose of 100 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 5 (Experimental): 4 Subjects will receive one dose of 200 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 6 (Experimental): 4 Subjects will receive one dose of 300 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 7 (Experimental): 4 Subjects will receive one dose of 400 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 8 (Experimental): 4 Subjects will receive one dose of 800 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 9 (Experimental): 4 Subjects will receive one dose of 1200 mg and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Single Ascending Dose Level 10 (Experimental): 4 Subjects will receive one dose on the outcome of preceding dose levels and 2 subjects will receive one dose of placebo
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 1 (Experimental): 6 Subjects will receive one dose of 50 mg each day for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose).
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 2 (Experimental): 6 Subjects will receive one dose of 200 mg each day for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 3 (Experimental): 6 Subjects will receive one dose of 400 mg each day for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 4 (Experimental): 6 Subjects will receive one dose of 800 mg each day for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 5 (Experimental): 6 Subjects will receive one dose of 1200 mg each day for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 6 (Experimental): 6 Subjects will receive one dose of 1200 mg each day (using tablet formulation instead of capsule formulation*) for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  *Tablet formulation is utilized, instead of capsule formulation, in the marked dose levels.
  Interventions: Drug: SKL24741; Drug: Placebo
- Food Effect Cohort (Experimental): After completing the fasting Single Ascending Dose escalation, the same 6 subjects who received one dose of 50 mg under fasting conditions will return to the clinic after a washout period for a second confinement to receive a second dose (same as fasting) under fed conditions.
  Interventions: Drug: SKL24741
- Gender Effect Cohort (Experimental): 6 female subjects of non-childbearing potential will receive one dose of 50 mg under fasting conditions.
  Interventions: Drug: SKL24741
- Optional Food Effect Cohort (Experimental): Up to 12 male subjects will undergo an open-label, two period, two-sequence crossover design at the maximum daily dose tested in Part A.
  Interventions: Drug: SKL24741
- Optional Formulation Effect Cohort (Experimental): Up to 12 male subjects will be treated with the maximum daily dose tested in Part A using open-label, two period, two-sequence crossover design.
  Interventions: Drug: SKL24741
- Multiple Ascending Dose Level 7 (Experimental): 6 Subjects will receive one dose of 2000 mg each day (using tablet formulation instead of capsule formulation*) for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  *Tablet formulation is utilized, instead of capsule formulation, in the marked dose levels.
  Interventions: Drug: SKL24741; Drug: Placebo
- Multiple Ascending Dose Level 8 (Experimental): 6 Subjects will receive one dose each day (using tablet formulation instead of capsule formulation*) for 14 days and 2 subjects will receive one dose placebo every day for 14 days. The dose will be determined based on the outcome of Part A (Single Ascending Dose) and/or preceding dose levels of Part B (Multiple Ascending Dose).
  *Tablet formulation is utilized, instead of capsule formulation, in the marked dose levels.
  Interventions: Drug: SKL24741; Drug: Placebo

INTERVENTIONS:
Drug: SKL24741 — An inhibitor of voltage-gated sodium channels and a possible activator of Big Potassium channels. Administered as an oral dose in the form of a capsule or tablet.
Drug: Placebo — Sugar pill manufactured to mimic SKL24741
  Arms: Multiple Ascending Dose Level 1; Multiple Ascending Dose Level 2; Multiple Ascending Dose Level 3; Multiple Ascending Dose Level 4; Multiple Ascending Dose Level 5; Multiple Ascending Dose Level 6; Multiple Ascending Dose Level 7; Multiple Ascending Dose Level 8; Single Ascending Dose Level 1; Single Ascending Dose Level 10; Single Ascending Dose Level 2; Single Ascending Dose Level 3; Single Ascending Dose Level 4; Single Ascending Dose Level 5; Single Ascending Dose Level 6; Single Ascending Dose Level 7; Single Ascending Dose Level 8; Single Ascending Dose Level 9

SUMMARY:
This study evaluates SKL24741 safety and tolerability in healthy subjects. Subjects will be randomized to receive oral doses of SKL24741 or placebo. This is a two-part, double-blinded, randomized study of SKL24741.

DETAILED DESCRIPTION:
The study includes a sequential cohort design that is intended to optimize subject safety and assess tolerability, safety, and PK of SKL24741. In the single-dose escalation part of the study (Part A), tolerability, safety, and PK of SKL24741 will be assessed in healthy male subjects under fasting conditions. At an appropriate dose based on PK results, additional cohorts will be repeated with the subjects under fed conditions, in order to evaluate the magnitude on the disposition of SKL24741. To assess the gender effect on the disposition of SKL24741, female subjects will be treated at one dose level under fasting conditions. A preliminary formulation effect may be assessed in a cohort of subjects to compare the capsule versus tablet formulation on the disposition of SKL24741.

Part A Primary Objective: To evaluate the safety and tolerability of single oral ascending doses of SKL24741 administered to healthy male subjects

Part A Secondary Objectives:

* To evaluate the PK of SKL24741 (R-enantiomer), SKL24742 (S-enantiomer) (if appropriate), and its possible metabolites (if deemed necessary) following administration of single oral ascending doses of SKL24741 administered to healthy male subjects
* To assess the food effect on the PK of SKL24741 and SKL24742 (if appropriate) following administration of a single oral dose of SKL24741 administered to healthy male subjects
* To assess the gender effect on the PK of SKL24741 and SKL24742 (if appropriate) following administration of a single oral dose of SKL24741 administered to healthy female subjects

Part A Exploratory Objective: To assess the formulation effect on the PK of SKL24741 and SKL24742 (if appropriate) following administration of a single oral dose of SKL24741 administered to healthy male subjects

Part B Primary Objective: To evaluate safety and tolerability of multiple oral ascending doses of SKL24741 administered for 14 days to healthy male subjects

Part B Secondary Objective: To evaluate the PK of SKL24741, SKL24742 (if appropriate), and its possible metabolites (if deemed necessary) following administration of multiple oral ascending doses of SKL24741 administered to healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects of 18 to 50 years of age (inclusive) except for the gender effect cohort
2. Able to read, understand, sign, and date a written informed consent form (ICF) before study participation at screening
3. Agree to use 2 highly effective methods of contraception, including at least one barrier method (Section 10.6.7 for details)
4. Body mass index (BMI) between 18.0 and 30.0 kg/m2 (inclusive) at screening
5. Judged to be in good health on the basis of medical history, physical examination, and routine laboratory measurements (i.e., without clinically relevant pathology)
6. Normal electrocardiogram (ECG) (12-lead), arterial blood pressure, and heart rate within the normal range of the study center or considered not clinically significant by the investigator and in agreement with the Sponsor
7. Able to understand and comply with protocol requirements and instructions and likely to complete the study as planned
8. For Part A (gender effect cohort): Female of non-childbearing potential (18 to 50 years of age (inclusive)), who have undergone a sterilization procedure at least 6 months prior to dosing with official documentation (e.g., hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy, hysterectomy, or bilateral oophorectomy), or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Principal Investigator's judgment

Exclusion Criteria:

1. History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subjects.
2. Smokers (subjects who have smoked within 6 months at screening or those with positive results from smoking screening).
3. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with pharmacokinetics of the trial medication (except appendectomy and simple hernia repair).
4. Regular treatment with prescription medications. Subjects should have ended any prescription medications at least 14 days before the first dosing of the study drug. Potential subjects should only stop any prescribed medication at the direction of a physician.
5. Regular treatment with nonprescription medications. Subjects should have ended any nonprescription medications at least 14 days before the first dosing of the study drug. Potential subjects should consult a physician before stopping any regular treatment with nonprescription medication.
6. Consumption of herbal medications, dietary supplements, and specific fruit products. Subjects should have stopped consumption of herbal medications or dietary supplements (e.g., St. John's Wort, ginkgo biloba, and garlic supplements), vitamins, and grapefruit or grapefruit juice, or Seville oranges at least 14 days before the first dosing of study drug.
7. History of drug or alcohol abuse or addiction within 2 years before the start of study drug dosing, or a positive test results for alcohol or drugs of abuse, such as amphetamine, barbiturate, benzodiazepine, cocaine, methadone, opiates, oxycodone, phencyclidine, propoxyphene, cannabinoid (THC), MDMA (Ecstasy), methaqualone, and tricyclic antidepressant (TCA).
8. Regular consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 pint [473 mL] of beer or lager, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) before screening. Subjects may not consume any alcohol from 72 hours before the first dosing of study drug through the completion of the last PK sampling.
9. Consumption of an average of more than 5 servings (8 ounces per serving) per day of coffee, cola, or other caffeinated beverage before screening. Subjects may not consume any caffeinated beverages from 48 hours prior to dosing until the collection of the last PK sample.
10. Participation in a clinical study involving administration of either an investigational or a marketed drug within 2 months or 7 half-lives (whichever is longer) before screening.
11. Blood donation or a significant loss of blood within 60 days of the start of study drug dosing or donation of more than 1 unit of plasma within 7 days before screening.
12. Positive result at screening for any of the following infectious disease tests: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antigen and antibody (HIV Ag, HIV Ab)
13. Illness within 5 days before the start of study drug dosing ("illness" is defined as an acute [serious or non-serious] condition [e.g., the flu or the common cold])
14. History of any known relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
15. Subject who is judged not eligible for study participation by investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will enroll up to 138 Healthy Male Subjects and 6 Non-childbearing potential Female Subjects.
Enrollment: 111 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Adverse events (Incidence of treatment-emergent adverse events) | From Screening until follow-up (14-16 days after dosing day or final dosing day)
  The number [count] and percentage [%] of subjects experiencing an adverse event
Clinically significant laboratory assessments | From Screening until follow-up (14-16 days after dosing day or final dosing day)
  Hematology, coagulation, clinical chemistry, urinalysis, and cholesterol
Electrocardiogram outcomes | From Screening until follow-up, including time-point assessments (In Part A, pre-dose until 24 hours post-dose. In Part B, Day1: pre-dose until 8 hours post-dose; Day 2-13: pre-dose only; Day 14: pre-dose until 24 hours post-dose)
  Standard electrocardiograms (ECGs) parameters will be measured, including heart rate (HR) [beats/min], RR [millisecond], PR [millisecond], QT [millisecond], QTc intervals [millisecond], and QRS duration [millisecond]. Extensive triplicate 12-lead ECGs, except for the food effect cohort, will be collected at various time points.
Vital sign | From Screening until follow-up, including time-point assessments (In Part A, Day1: pre-dose until 12 hours post-dose. In Part B, Day1: pre-dose until 12 hours post-dose; Day 2-14: pre-dose until 8 hours post-dose)
  Blood pressure (systolic and diastolic measurements in supine and standing in the same sequence in each subject, in order to allow orthostatic measurements) [mmHg]
Vital sign | From Screening until follow-up, including time-point assessments (In Part A, Day1: pre-dose until 12 hours post-dose. In Part B, Day1: pre-dose until 12 hours post-dose; Day 2-14: pre-dose until 8 hours post-dose)
  Temperature [Celsius]
Vital sign | From Screening until follow-up, including time-point assessments (In Part A, Day1: pre-dose until 12 hours post-dose. In Part B, Day1: pre-dose until 12 hours post-dose; Day 2-14: pre-dose until 8 hours post-dose)
  Heart rate [beats/min]
Vital sign | From Screening until follow-up, including time-point assessments (In Part A, Day1: pre-dose until 12 hours post-dose. In Part B, Day1: pre-dose until 12 hours post-dose; Day 2-14: pre-dose until 8 hours post-dose)
  Respiratory rate [breaths/min]
Vital signs | From Screening until follow-up, including time-point assessments (In Part A, Day1: pre-dose until 12 hours post-dose. In Part B, Day1: pre-dose until 12 hours post-dose; Day 2-14: pre-dose until 8 hours post-dose)
  Arterial oxygen saturation (SaO2) (using pulse oximetry) [%]
Physical examination | Full (complete) physical examination at screening only. From Screening until follow-up (14-16 days after dosing day or final dosing day)
  Full physical examination (review of all body systems - head/neck/thyroid, eyes/ears/nose/throat, respiratory, cardiovascular, lymph nodes, abdomen, skin, musculoskeletal, and neurological. Breast, anorectal, and genital examinations)
Physical examination | Full (complete) physical examination at screening only. From Screening until follow-up (14-16 days after dosing day or final dosing day)
  Height [centimeter]
Physical examination | Full (complete) physical examination at screening only. From Screening until follow-up (14-16 days after dosing day or final dosing day)
  Weight [kg]
Physical examination | Full (complete) physical examination at screening only. From Screening until follow-up (14-16 days after dosing day or final dosing day)
  BMI [kg/m^2]
Physical examination | Full (complete) physical examination at screening only. From Screening until follow-up (14-16 days after dosing day or final dosing day)
  Abbreviated (symptom-directed) physical examination.
Peak expiratory flow rate | Assessed at admission (Day -1), pre-dose (baseline), 2 and 24 hours post-dose after the first dose (Day 1 dosing) and the last dose (Day 14 dosing for Part B), and follow-up (14-16 days after dosing day or final dosing day)
  Peak expiratory flow rate [L/min], the maximum rate that a person can exhale during a short maximal expiratory effort after a full inspiration
Columbia-Suicide Severity Rating Scale (Part B only) | From Screening until follow-up (14-16 days after dosing day or final dosing day). Baseline ("Lifetime/Recent") at Screening and "Since Last Visit" versions on other visits
  Columbia-Suicide Severity Rating Scale (C-SSRS) is a brief questionnaire that provides for the identification, quantification, and standardized assessment of the occurrences and severity of suicidal ideation and behavior. The changes from baseline and clinical abnormalities will be assessed (units on a scale).

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Maximum concentration (Cmax) [ng/mL] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Time to maximum concentration (tmax) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Time to maximum concentration (tmax) [hours, or h] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Area under the concentration-time curve (AUC) from 0 to infinity (AUC∞) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Area under the concentration-time curve (AUC) from 0 to infinity (AUC∞) [ng*h/mL] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles after a single dose administration
AUC from time 0 to a given time t (AUCt) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  AUC from time 0 to a given time t (AUCt) [ng*h/mL] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
AUC over the dosing interval (AUCτ) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  AUC over the dosing interval (AUCτ) [ng*h/mL] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Apparent clearance (CL/F) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Apparent clearance (CL/F) [L/h] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Apparent volume of distribution (Vd/F) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Apparent volume of distribution (Vd/F) [Liter, or L] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Half-life (t1/2) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Half-life (t1/2) [hour] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles
Accumulation ratio (Racc) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single and/or multiple dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose plasma samples. In Part B, Days 1 and 7: pre-dose and up to 24 hours post-dose, Days 3-6 and 9-13: pre-dose only, and Day 14: Pre-dose and up to 240 hours post-dose plasma samples
  Accumulation ratio (Racc) [unit of ratio] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the plasma concentration-time profiles

OTHER OUTCOMES:
Fraction excreted unchanged in the urine (fe) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose urine samples.
  Fraction excreted unchanged in the urine (fe) [unit of fraction] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the urine concentration-time profiles
Renal clearance (CLr) of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) following the single dose administration of SKL24741 | In Part A, pre-dose and up to 240 hours post-dose urine samples.
  Renal clearance (CLr) [Liter/h or milliliter/min] of SKL24741, SKL24742 (if appropriate), and possible metabolites (if deemed necessary) for the urine concentration-time profiles

CONTACTS AND LOCATIONS:
Overall Officials: Vijaykumar Vashi, PhD, Study Director — SK Life Science, Inc.
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT04505397/Prot_000.pdf